CLINICAL TRIAL: NCT00941902
Title: A Potential Novel Marker for Liver Fibrosis in Nonalcoholic Steatohepatitis: the Soluble Secreted Form of the Human Asialoglycoprotein Receptor Non-interventional Study.
Brief Title: A Potential Novel Marker for Liver Fibrosis in NASH: the Soluble Secreted Form of the Human Asialoglycoprotein Receptor
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Dr. Hussein Osamah, Ziv Medical Center
Other Study IDs: 0022-09 ZIV
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Liver Fibrosis
Keywords: human asialoglycoprotein receptor (ASGPR); hepatocytes; bariatric surgery
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients scheduled to bariatric surgery

SUMMARY:
Soluble secreted proteins that are expressed uniquely in specific organs and whose formation of secretion is regulated by disease states are excellent markers for the disease. This is because the disease can be diagnosed by simply measuring the levels of the secreted protein in serum. A soluble form of the asialoglycoprotein receptor could be a promising candidate for such marker in the case of liver fibrosis secondary to steatohepatitis for which the existing markers are not satisfactory. The human asialoglycoprotein receptor (ASGPR) is expressed only in hepatocytes. The H2a alternatively spliced variant of the ASGPR H2 subunit differs from H2b variant only by the presence of an extra pentapeptide. EGHRG, in the exoplasmic domain next to the membrane-spanning segment. H2a is rapidly cleaved to a36 kDa fragment, comprising the entire ectodomain, which is secreted. H2a does not participate in a membrane bound receptor complex with H1 as in the case for H2b and thus it is not a subunit of the receptor but a precursor for a soluble secreted form of the protein (sH2a). Although H2a is a type II transmembrane protein, signal peptidase is probably responsible for the cleavage to the soluble form.

The objective in this research proposal is to study the association between the level of sH2a. in the serum and the severity of fibrosis in steatohepatitis in patients undergoing bariatric surgery due to morbid obesity.

The existence of sH2a in normal human serum is at very constant levels. On the other hand the membrane ASGPR (expressed exclusively in hepatocytes) is profoundly down - regulated in liver cancer and cirrhosis. The investigators will analyze the levels of sH2a in serum from patients with steatohepatitis in different stages of fibrosis and compare with healthy subjects. A possible early down-regulation of sH2a in fibrosis may prove to be a valuable diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Patient candidate to bariatric surgery.

Exclusion Criteria:

1. Liver biopsy during the last 12 months.
2. The surgeon consider liver biopsy as a special dander in a specific patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to bariatric surgery will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Hussein, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- ZIV Medical Center, Safed, Israel